CLINICAL TRIAL: NCT00275977
Title: Treatment of Myocardial Infarction With Autologous Bone Marrow Derived Stem Cells
Brief Title: Treatment of Myocardial Infarction With Bone Marrow Derived Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 020
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2006-01

CONDITIONS: Acute Myocardial Infarction
Keywords: "Stem cell"; "autologous bone marrow transplantation"; "Myocardial infarction"
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Procedure: Coronary catherization and stem cell infusion

SUMMARY:
The aim of the study is to investigate whether infusion of autologous bone marrow derived stem cells can improve cardiac function in the aftermath of a myocardial infarction.

DETAILED DESCRIPTION:
Primary coronary intervention within a few hours of a myocardial infarction has greatly reduced mortality as well as the risk of developing chronic heart failure. There are though still a large number of patients that develop symptoms of heart failure in the form of fatigue and breathlessness with physical exertion in spite of medical treatment. With the advance in stem cell technology there is now hope for the possibility of regenerating/repairing dead myocardial tissue, hence improving cardiac function.

The current study is a pilot study that is going to precede a later double blinded randomized study. The aim of the study is to evaluate patient safety, optimize procedures, and to be used in power calculation in the design of the following study.

ELIGIBILITY:
Inclusion Criteria:

* Chestpain
* Troponin T, > 0,1ng/ml
* Succesfull revascularization of culprit lesion with PCI.
* No more than stenosis of 2 major epicardiel coronary arteries.

Exclusion Criteria:

* Cardiogenic shock
* Known LVEF<45%
* Cardiomyopathy
* Atrialfibrillation or fluctuation
* Takyarytmia
* Infection
* Chronic inflammatory disease

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-02; Study Completion 2007-03

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Change in left ventricular funtion at 4 months followup using contrast enhanced echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha Kassem, MD, Ph.D, Principal Investigator — Department of endocrinology M, Odense University Hospital
Locations (1):
- Department of endocrinology M, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Wollert KC, Meyer GP, Lotz J, Ringes-Lichtenberg S, Lippolt P, Breidenbach C, Fichtner S, Korte T, Hornig B, Messinger D, Arseniev L, Hertenstein B, Ganser A, Drexler H. Intracoronary autologous bone-marrow cell transfer after myocardial infarction: the BOOST randomised controlled clinical trial. Lancet. 2004 Jul 10-16;364(9429):141-8. doi: 10.1016/S0140-6736(04)16626-9. PMID 15246726
- [Background] Schachinger V, Assmus B, Britten MB, Honold J, Lehmann R, Teupe C, Abolmaali ND, Vogl TJ, Hofmann WK, Martin H, Dimmeler S, Zeiher AM. Transplantation of progenitor cells and regeneration enhancement in acute myocardial infarction: final one-year results of the TOPCARE-AMI Trial. J Am Coll Cardiol. 2004 Oct 19;44(8):1690-9. doi: 10.1016/j.jacc.2004.08.014. PMID 15489105